CLINICAL TRIAL: NCT05896540
Title: Study Protocol: a Randomized Controlled Trial of a Gender-transformative School-based Sexual Health Intervention in Chilean Students
Brief Title: Randomized Controlled Trial of a Gender-transformative School-based Sexual Health Intervention
Acronym: ENFOCATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Chile (Other)
Collaborators: National Fund for Research and Development in Health, Chile (Other)
Responsible Party: Principal Investigator, Loreto Leiva, Associate professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FONIS SA21I0142
Record Dates: First submitted 2023-01-30; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Sexuality
Keywords: School-based sexual health intervention; Gender perspective; School intervention
MeSH Terms: conditions — Sexuality

STUDY DESIGN:
Intervention Model Description: The assignment of the participants to the groups will be implemented in a two-stage selection of the students; since there are already existing teaching-learning processes in process in the schools, with their time limitations, the investigators will have to choose entire "courses" (in Chilean secondary schools, a course is a group of about 40 students who have all classes together) rather than choose individual students. The investigators will establish groups among the schools to compensate for their different sizes; some schools in the commune are much larger than the others (four or more courses per grade. Thus the investigators will divide the schools into two blocks; one with the largest schools and one with the medium- and small-sized schools. In the second stage, courses that meet the inclusion criteria to participate in the study will be selected randomly within each of the blocks. Table 1 details the distribution of the samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STUDY GROUP ENFOCATE (Experimental): The selected students will be randomly divided into the study and control groups; the intervention will take place in the same schools that the students attend. The assignment to groups will use simple random sampling, performed in two stages. In the first stage the available schools will be randomly assigned to the study and control groups, while the second stage will select randomly the groups in each school that will participate in the study. The study groups will receive a 10-session intervention in sexual education, covering topics related to preventive sexual conduct, gender equity and mental health.
  Interventions: Behavioral: ENFOCATE
- CONTROL GROUP (No Intervention): The control groups will not receive intervention; they will continue with the sexual orientation that each school provides to its students.

INTERVENTIONS:
Behavioral: ENFOCATE — ENFOCATE is a comprehensive program of sexual education for adolescents. Its design follows the guidelines of the Intervention Mapping Approach and the orientations proposed by the Framework for Gender-Transformative Health Promotion. The intervention has a participative focus, thus the activities are designed to promote processes of knowledge, understanding, application and reflection in the adolescents. The activities aim to improve the capacity for critical thinking, increase the motivation to listen and learn actively, and to improve interpersonal abilities. The execution of the intervention uses three pillars: (i) preventive sexual behavior; (ii) gender equity; and (iii) mental health. The intervention consists of ten weekly sessions, each lasting one hour. The teams that will perform the intervention will be composed of at least two professionals of the psychosocial area (mainly psychologists, social workers and/or guidance counsellors) of the schools included in the study.
  Arms: STUDY GROUP ENFOCATE

SUMMARY:
The goal of this randomized controlled trial (RCT) is to evaluate the effectiveness of a comprehensive gender-transformative intervention of sexual education (ENFOCATE -Focus-on) in adolescents, using a mixed experimental design. The intervention will be directed exclusively to students of the 10th and 11th grades who are enrolled in one of the education establishments that depend on the Municipality of Santiago. The randomization will be by grade, and the data will be collected at three moments (pre-intervention, post-intervention and a 3-month follow-up).

DETAILED DESCRIPTION:
The investigators propose a mixed experimental design with a randomized controlled trial (RCT) that will evaluate the efficiency of an intervention and implementation of a comprehensive gender-transformative sexual education, along with qualitative studies to understand the implementation process. The results of the intervention will be evaluated after it finishes, and in a three-month follow-up. Each participant will be sent a link to the questionnaire (web-based survey). Follow-up contact will be done with WhatsApp or telephone calls.

The hypothesis is that the intervention designed and implemented in the experimental group: (1) will increase their sexuality knowledge level; (2) will increase their preventive sexual behavior (or intentions); (3) will favor a gender-positive attitude; and (4) will decrease internalizing and externalizing problems in mental health. The secondary objective is to examine the implementation intervention process, that is, identify the strengths and obstacles in the real context in which the study intervention is performed, to understand the determinants and strategies of the success of the implementation.

ELIGIBILITY:
Inclusion Criteria

* Schools with students of the 10th and 11th grades who are enrolled in one of the education establishments that depend on the Municipality of Santiago.
* Schools not being an education center oriented to adults or persons deprived of liberty (e.g. closed or semi-closed compounds of Gendarmería de Chile or the National Service for Minors)
* Schools with regularity in teaching and learning (for example, schools that were not partially interrupted in 2022 by student manifestations)
* Schools with informed consent of the director.
* Students having 90% or greater attendance in classes
* Students providing informed consent of voluntary participation
* Students having explicit and informed consent of their parents or guardians.

Exclusion Criteria:

* Schools being an education center oriented to adults or persons deprived of liberty
* Schools without informed consent of the director
* Students without class attendance
* Students without informed consent of voluntary participation
* Students without an explicit and informed consent of their parents or guardians

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 609 (Estimated)
Dates: Start 2023-08-05 (Estimated); Primary Completion 2023-09-03 (Estimated); Study Completion 2023-12-29 (Estimated)

PRIMARY OUTCOMES:
Change in knowledge of sexuality | One-week pre-intervention, immediately post-intervention and a 3-month follow-up
  Related to information about the biological components of sexuality. The test used will be the Knowledge Test (KT). This is a 34-item multiple choice instrument which was designed to evaluate the knowledge on sexuality in adolescents; it evaluates areas including pregnancy, STI, physical development. Higher scores represent more favorable attitudes. Its reliability is α=0.89. These assessed areas will be combined to report the level of knowledge.
Change in preventive sexual behavior | One-week pre-intervention, immediately post-intervention and a 3-month follow-up
  Related to behavior in sexuality and preventive behavior in sexuality. Ad-hoc survey. It will be elaborated by the research team to evaluate the behavior and intention, self-efficacy and empowerment in sexuality in LGTB and female-male students. Ad-hoc surveys have been used and reported in other RCT of interventions in sexual health.
Change in gender actitude | One-week pre-intervention, immediately post-intervention and a 3-month follow-up
  Related to positive disposition towards persons of different genders. The test used will be the Scale for Detection of Sexism in adolescents (DSA). This is an instrument of 26 items developed for adolescents. It evaluates sexism, differentiating between hostile and benevolent sexism. The response scale for the items is a Likert type with six alternatives (from 1=disagree completely to 6=agree completely). Higher scores indicate more sexism. Its reliability is α= .881.
Change in gender actitude | One-week pre-intervention, immediately post-intervention and a 3-month follow-up
  Related to positive disposition towards persons of different sexual orientation. The test used will be the Scale of negative attitudes toward trans persons (NATP). It measures attitude as an expression of prejudice towards trans persons. It has nine items with a Likert scale with five response options, from 1= disagree completely to 5=agree completely. Higher scores are indicators of higher levels of negative attitudes toward persons of different sexual orientation. Its reliability is α= .886.
Change in gender actitude | One-week pre-intervention, immediately post-intervention and a 3-month follow-up
  Related to positive disposition towards persons of different sexual orientation. The test used will be the Short version of Modern Homophobia Scale (MHS). It measures homophobic attitudes in the dimension personal discomfort, institutional and deviation/changeability. It is composed of 46 items that evaluate attitudes towards lesbians and gay in a Likert scale of 1-5 in which higher scores interpret more positive attitudes towards homosexuality and lesbianism. Its reliability is α= .80.
Change in components of mental health related to sexual health | One-week pre-intervention, immediately post-intervention and a 3-month follow-up
  Decrease of internalizing symptomology. The test used will be the Pediatric Symptom Checklist (PSC-17). It evaluates general psychosocial functioning, detecting emotional and behavioral difficulties in children and adolescents. Higher scores represent more internalizing behaviors. reliability is α= .72.
Change in components of mental health related to sexual health | One-week pre-intervention, immediately post-intervention and a 3-month follow-up
  Decrease of externalizing symptomology. The test used will be the Pediatric Symptom Checklist (PSC-17). It evaluates general psychosocial functioning, detecting emotional and behavioral difficulties in children and adolescents. Higher scores represent more externalizing behaviors. Its reliability is α= .72.

CONTACTS AND LOCATIONS:
Overall Officials: Loreto Leiva, PhD, Principal Investigator — University of Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leiva L, Torres-Cortes B, Antivilo-Bruna A, Zavala-Villalon G. Gender-transformative school-based sexual health intervention: study protocol for a randomized controlled trial. Trials. 2024 Jun 5;25(1):360. doi: 10.1186/s13063-024-08191-w. PMID 38835035